CLINICAL TRIAL: NCT04084639
Title: To Determine the Effects of Mycoprotein Consumption on Glucose Absorption in Healthy Participants
Brief Title: Mycoprotein Consumption and Glucose Absorption
Acronym: MEGA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: Quorn (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 190206/B/06
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind crossover design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ingestion of 20g Mycoprotein Drink (Experimental): Milkshake containing 20g of mycoprotein, 250ml full-fat milk, 50g glucose and 11g lactose is given to participants in one dose
  Interventions: Dietary Supplement: Mycoprotein Ingestion
- Ingestion of 40g Mycoprotein Drink (Experimental): Milkshake containing 40g of mycoprotein, 250ml full-fat milk, 50g glucose and 11g lactose is given to participants in one dose
  Interventions: Dietary Supplement: Mycoprotein Ingestion
- Ingestion of Isocaloric Control Drink (Placebo Comparator): Milkshake containing 250ml full-fat milk, 50g glucose, 19g dried skim milk and 9g full-fat dried milk
  Interventions: Dietary Supplement: Mycoprotein Ingestion

INTERVENTIONS:
Dietary Supplement: Mycoprotein Ingestion — Ingestion of various doses of mycoprotein compared to placebo control

SUMMARY:
Previous research has demonstrated that the food found in Quorn 'Mycoprotein' can lower the blood glucose response to a meal, which may be an important finding for the management of type 2 diabetes. However, it has never been investigated how this lower response occurs, and whether there is dose-dependent response with mycoprotein. The present study will include 12 healthy young adults, who will visit the laboratory for 3 test days, with each day lasting 9 hours. On each visit, separated by a washout period of at least 2 weeks, participants will ingest either a control drink with no mycoprotein, a drink containing 20g mycoprotein or a drink containing 40g mycoprotein. By intravenously infusing labelled glucose during each visit in combination with repeated blood sampling, investigators will determine if the lower blood glucose after mycoprotein ingestion is due to reduced glucose absorption from the gut or increased uptake into body tissues.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* 18-35 years of age
* Consumption of sufficient amounts of carbohydrate in the diet
* Body mass index between 18.5 and 30

Exclusion Criteria:

* Any diagnosed metabolic impairment (e.g. type 1 or 2 Diabetes), or other form of abnormal glucose metabolism (as this will affect outcome of the study).
* Any diagnosed cardiovascular disease
* Insufficient consumption of carbohydrate in the diet
* A personal or family history of epilepsy, seizures or schizophrenia
* Known pre-existing liver disease/condition
* Allergy or intolerance to milk

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
Glucose absorption | 6 hours following ingestion of drink
  How glucose is absorbed following the ingestion of a mycoprotein drink compared to a placebo control measured using the infusion of stable isotopes

SECONDARY OUTCOMES:
Incretin Hormones | 6 hours following ingestion of drink
  Measurement of glucagon-like peptide-1(GLP-1) and gastric inhibitory polypeptide (GIP) in response to mycoprotein ingestion compared to placebo control
Insulinaemic Response | 6 hours following ingestion of drink
  Measurement of insulin response following ingestion of drinks
Production of Short-Chain Fatty Acids | 6 hours following ingestion of drink
  Measurement of plasma acetate production in response to mycoprotein ingestion
Glucose Kinetics | 6 hours following ingestion of drink
  Calculations using plasma deuterated glucose enrichment to determine rate of appearance of endogenous glucose, rate of disappearance of glucose and rate of appearance of exogenous glucose

CONTACTS AND LOCATIONS:
Locations (1):
- University of Exeter, Exeter, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Whelehan G, West S, Abdelrahman DR, Murton AJ, Finnigan TJA, Wall BT, Stephens FB. The addition of mycoprotein to a mixed-meal impacts postprandial glucose kinetics without altering blood glucose concentrations: a randomised controlled trial. Eur J Clin Nutr. 2024 Sep;78(9):757-764. doi: 10.1038/s41430-024-01470-4. Epub 2024 Jul 13. PMID 39003347